CLINICAL TRIAL: NCT06390501
Title: The Effect of Weekly Semaglutide Treatment on Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Chief Scientist, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SIAT-IRB-231215-H0705
Record Dates: First submitted 2024-04-11; First posted 2024-04-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Drug
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Once-weekly injections of gradually increased doses of semaglutide
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Once-weekly injections of gradually increased volumes of saline placebo, to match the volumes of the semaglutide treated arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Solution for subcutaneous (s.c. - under the skin) injection. 0.25 mg semaglutide once weekly for four weeks, 0.5 mg semaglutide once weekly for four weeks, 0.1 mg semaglutide once weekly for four weeks, 1.7 mg semaglutide once weekly for four weeks followed by 2.4 mg semaglutide once weekly for eight weeks
  Arms: Semaglutide
Drug: Placebo — Solution for subcutaneous (s.c. - under the skin) injection
  Arms: Placebo

SUMMARY:
This study will test the effects of weekly injections of the glucagon like peptide-1 (GLP-1) agonist semaglutide on energy expenditure and metabolic parameters in a 24 week double-blind, placebo-controlled dose escalation randomized trial. After baseline testing, 52 patients will be randomly assigned to the semaglutide or matching placebo injection group. In addition to taking medication or placebo, all participants will a calorie restricted diet provided by the researchers, providing 600 kcals per day below their estimated baseline requirements. Before and at the end of treatment, weight status, body composition, basal metabolic rate (BEE), 24h energy expenditure, daily total energy expenditure (TEE) for free living, physical activity, energy intake (questionnaire and food table), and hormone parameters for energy homeostasis will be evaluated.

DETAILED DESCRIPTION:
Obesity is a complex chronic recurrent multifactorial disease characterized by abnormal or excessive body fat, which impairs physical health. In recent years, the glucagon like peptide-1 (GLP-1) receptor agonist semaglutide has attracted much attention due to its significant impact on weight loss. It can not only effectively control blood sugar by regulating the secretion of insulin and glucagon. It can also participate in certain brain regions of the body at pharmacological doses, regulating food intake and consumption. Semaglutide reduces energy intake and achieves weight loss by delaying gastric emptying, suppressing appetite, reducing hunger, and increasing satiety. This effect has been proven to be produced by activating the glucagon like peptide-1 (GLP-1) receptors in the central nervous system, further indirectly regulating the activity of neurons involved in appetite regulation, food intake, and preference.

The previous results of using GLP-1 receptor agonist (RA) in rats and humans provide promising evidence data to support current randomized clinical trials. Peripheral administration of GLP-1 or GLP-1 RA can reduce blood sugar and energy intake in humans and rodents, and long-term treatment can lead to weight loss. In mice the drug also sustains energy expenditure at levels similar to controls, preventing the reduction that normally accompanies caloric restriction. Whether the same effects occur in humans is unclear because no studies have yet been performed comparing semaglutide treated individuals with those on a standard calorie restricted diet (in effect pair feeding). Therefore, in this study, researchers will use doubly- labelled water (DLW) and respiratory chambers to investigate whether semaglutide can prevent the reduction of energy expenditure that typically occurs during energy restriction.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-60 years at time of enrollment
2. BMI ≥ 25 kg/m²

Exclusion criteria:

1. Weight change exceeding 5 kilograms (11 pounds) in the past 90 days
2. Surgical treatment for past obesity, dieting, or undergoing weight loss treatment
3. Irregular diet and lifestyle, unhealthy habits such as smoking, alcohol, and drugs
4. Patients with metabolic diseases, basic diseases or infectious diseases
5. Patients with a personal or family history of medullary thyroid carcinoma (MTC), or patients with rare type 2 multiple endocrine tumor syndrome (MEN 2)
6. Current use of any other GLP1 receptor agonist
7. Pregnancy, lactation or expectation to conceive during study period (8) Subject with contraindication to neuroimaging by MRI (9) People with fear of blood and pathologically low blood pressure (10) Use of antibiotics and probiotics within 8 weeks

11) Subject unlikely to adhere to study procedures in opinion of investigator

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Changes of Total Energy Expenditure Assessed by Doubly Labeled Water Analysis | From baseline at week 0 to week 24
  TEE will be measured using the DLW method. Urine samples from all participants in the DLW subset will be stored at -20 ℃ and shipped on dry ice for analysis in the laboratory of Dr. John Speakman at the Shenzhen Institute of Advanced Technology, Chinese academy of sciences. Isotopes will be measured in benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation (Speakman et al 2021: Cell reports medicine). TEE will then be calculated using mean CO2 production using the Weir equation.
Changes of Energy Expenditure Assessed by Chamber | From baseline at week 0 to week 24
  The total energy expenditure in a free living environment is measured using a 24-hour chamber.
Changes of Resting Energy Expenditure | From baseline at week 0 to week 24
  Resting energy expenditure will be measured using indirect calorimetry via a respiratory hood system (Cosmed). The subject attends in the lab after an overnight fast. The person lies down on a flat bed and the hood is placed over their head. Metabolic rate (oxygen consumption and CO2 production) are monitored for 40 minutes. The last 10 minutes is used as the measurement. Calorimeters will be assessed with a turbine test to ensure accuracy of measurements. Validation via an alcohol burn will be performed monthly.
Changes of Physical Activity | From baseline at week 0 to week 24
  Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 14 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day where the wear time is less than 12 hours. For a valid measure the goal is to get 2 weekday and 2 weekend days.

SECONDARY OUTCOMES:
Body Weight | From baseline at week 0 to week 24
  Subjects will be asked to fast overnight and weight will be measured using a calibrated Seca body weight scale first thing in the morning on subjects wearing light clothes and no shoes.
Body Mass Index (BMI) | From baseline at week 0 to week 24
  Percent change of body mass index (BMI), as calculated by the formula: body weight in kg divided by height in meters², between baseline and the end of the 24-week randomized drug treatment phase.
Waist and Hip circumferences | From baseline at week 0 to week 24
  Waist and Hip circumferences will be measured using a whole body laser scanner.
Body shape | From baseline at week 0 to week 24
  Body shape will be measured using a whole body laser scanner.
Fat mass | From baseline at week 0 to week 24
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Far free mass | From baseline at week 0 to week 24
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980).
Organ sizes | From baseline at week 0 to week 24
  Volumes of the brain, liver, spleen, pancreas, kidneys, subcutaneous and visceral adipose tissue, skeletal muscle in the limbs, trunk and shoulders will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Bone mass | From baseline at week 0 to week 24
  Bone mass will be measured by Dual Energy X-ray Absorptiometry (DEXA) (Hologic)
Changes in Body Composition as Assessed by Body Fat Mass Using Dual Energy X-ray Absorptiometry (DEXA) | From baseline at week 0 to week 24
  Body composition change between baseline and the end of the 24-week randomized drug treatment phase assessed by dual energy x-ray absorptiometry (DEXA) and expressed as the change in fat mass.
Change in energy intake of test meal | From baseline at week 0 to week 24
  The food intake will be assessed objectively by use of a feeding table. The test meal will be provided as lunch, and food types available on the table include staples, vegetables, mushrooms, meat, soy products, desserts, beverages and water. All types of food are unlimited. Food consumption will be recorded continuously by balances concealed under each food dish. The food energy density for each food will be measured by bomb calorimetry in kJ/g, and energy intake will be calculated as the product of the grams of each food eaten multiplied by the respective energy density and then summed, as kJ.
Changes in Fat and Total Calorie Intake Assessed by Free Buffet Meal Analysis | From baseline at week 0 to week 24
  Changes in fat and total calorie intake during free buffet meals assessed at baseline and after 24-weeks of study drug treatment.
Energy intake during ad libitum lunch | From baseline at week 0 to week 24
  The food intake will be assessed objectively by use of a feeding table. The test meal will be provided as lunch, and food types available on the table include staples, vegetables, mushrooms, meat, soy products, desserts, beverages and water. All types of food are unlimited. Food consumption will be recorded continuously by balances concealed under each food dish. The food energy density for each food will be measured by bomb calorimetry in kJ/g, and energy intake will be calculated as the product of the grams of each food eaten multiplied by the respective energy density and then summed, as kJ.
Body temperature from surface temperature of the forehead | From baseline at week 0 to week 24
  Body temperature will be measured before and after feeding using a thermal imaging camera. The camera is directed at the forehead to measure the surface temperature.
Body water | From baseline at week 0 to week 24
  Body water will be measured by deuterium dilution. Subjects will attend in the lab after an overnight fast and provide a baseline urine sample. They will then drink a dose of deuterated water based on their body weight. Three and four hours after dosing a urine sample will be collected to measure the level of deuterium isotope in the body relative to the baseline. This increase allows measurement of the amount of water in the body that diluted the dose.
Overall appetite score (OAS) before and after intake of a standardised meal | From baseline at week 0 to week 24
  give a score from 0 to 100
Mean postprandial rating - Hunger | From baseline at week 0 to week 24
  give a score from 0 to 100, The ends of each line indicate the most extreme sensation respondents have experienced
Mean postprandial rating - Fullness | From baseline at week 0 to week 24
  give a score from 0 to 100, The ends of each line indicate the most extreme sensation respondents have experienced
Mean postprandial rating - Satiety | From baseline at week 0 to week 24
  give a score from 0 to 100, The ends of each line indicate the most extreme sensation respondents have experienced
Mean postprandial rating - Prospective food consumption | From baseline at week 0 to week 24
  give a score from 0 to 100, The ends of each line indicate the most extreme sensation respondents have experienced
Change in physical functioning score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: role-physical score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: bodily pain score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: general health score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: vitality score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: social functioning score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: role-emotional score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: mental health score | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: physical component summary | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Change in SF-36: mental component summary | From baseline at week 0 to week 24
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Subjects who achieve responder definition value for SF-36 physical functioning score (yes/no) | From baseline at week 0 to week 24
  Number of subjects
Change in HbA1c | From baseline at week 0 to week 24
  mmol /mol
Change in systolic and diastolic blood pressure | From baseline at week 0 to week 24
  Systolic and diastolic blood pressure will be measured using an Omron digital sphygmomanometer, as mmHg.
Blood glucose | From baseline at week 0 to week 24
  Fasting and post-prandial glucose after a standard meal will be recorded by a continuous glucose monitoring system.
Change in fasting serum insulin | From baseline at week 0 to week 24
  mIU/L
Change in lipids: Total cholesterol | From baseline at week 0 to week 24
  mg/dL
Change in lipids: High density lipoprotein (HDL) cholesterol | From baseline at week 0 to week 24
  mg/dL
Change in lipids: Low density lipoprotein (LDL) cholesterol | From baseline at week 0 to week 24
  mg/dL
Change in lipids: Very low density lipoprotein (VLDL) cholesterol | From baseline at week 0 to week 24
  mg/dL
Change in lipids: Free fatty acids (FFA) | From baseline at week 0 to week 24
  mg/dL
Change in lipids: Triglycerides | From baseline at week 0 to week 24
  mg/dL
Change in fatty liver index (FLI) score category | From baseline at week 0 to week 24
  Below 30, equal to or above 30 and below 60, equal to or above 60
Changes in Inflammation Assessed by C-reactive Protein (CRP) | From baseline at week 0 to week 24
  Change in C-reactive protein (CRP) between baseline and the end of the 24-week randomized drug treatment phase
Subjects who have permanently discontinued randomised trial product (yes/no) | From baseline at week 0 to week 24
  Number of subjects
Time to permanent discontinuation of randomised trial product | From baseline at week 0 to week 24
  Weeks
Number of treatment emergent adverse events (TEAEs) | From baseline at week 0 to week 24
  Count
Number of serious adverse events (SAEs) | From baseline at week 0 to week 24
  Count
Change in pulse | From baseline at week 0 to week 24
  Beats per minute (bpm)
Change in amylase | From baseline at week 0 to week 24
  U/L
Change in lipase | From baseline at week 0 to week 24
  U/L
Changes of Circulating Leptin Levels | From baseline at week 0 to week 24
  Change in circulating leptin between baseline and the end of the 24-week randomized drug treatment phase
Circulating hormones | From baseline at week 0 to week 24
  Nurses will collect the blood samples every month. Levels of circulating hormones (including leptin, insulin, ghrelin etc) and metabolic fuels (glycogen, lactate glucose etc) will be measured when fasted and after a standard intervention meal. Levels of circulating hormones in the serum will be measured by ELISA (Bio Tek, Synergy4) in mmol/L.
Microbiome | From baseline at week 0 to week 24
  Abundance of gut microbiome will be from Metagenomic profiling of feces by Illumina.
Metabolites in serum, feces and urine | From baseline at week 0 to week 24
  Abundance of metabolites will be from metabolomic profiling of serum, urine and feces by LC-MS (liquid chromatography-mass spectrometry).
Genetics | From baseline at week 0 to week 24
  Polymorphic variation will be assessed in a panel of SNPs (single nucleotide polymorphism) previously linked to body composition and physical activity using a Mass array sequencer.
  OR The subjects will have their venous blood collected in a fasted state. 4ml of venous blood (BD vacutainer K2 EDTA, BD, USA) will be used to extract genomic DNA (TIANamp Blood DNA kit, TIANGEN, China. QIAamp Midi Blood DNA kit, QIAGEN, Germany) for Single nucleotide polymorphism (SNP) genotyping (Agena MassARRAY, CapitalBio Technology, China).

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Shenzhen, China